CLINICAL TRIAL: NCT01487408
Title: Special Survey for Type 1 or Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-1944
Record Dates: First submitted 2011-11-29; First posted 2011-12-07 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin Aspart
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Adminstered subcutaneously (s.c., under the skin). Prescribed by physician as a results of normal clinical practice

SUMMARY:
This study is conducted in Japan. The aim of this study is to evaluate the incidence of severe hypoglycaemia episodes under normal clinical practice for patients with type 1 or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes requiring insulin therapy

Exclusion Criteria:

* Patients who had not been treated more than 3 months at the same investigational site
* Patients who had treatment history of NovoRapid® (insulin aspart)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 1 or type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 1463 (Actual)
Dates: Start 2002-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Incidence of servere hypoglycaemia
Total dose of insulin (aspart/human insulin) infused subcutaneously
Physical examination
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com